CLINICAL TRIAL: NCT06917404
Title: A Phase 3, Randomised, Double-Blind, Placebo-Controlled Multi-Centre Study to Evaluate the Treatment Effect of Pentosan Polysulfate Sodium Compared to Placebo in Participants With Knee Osteoarthritis Pain
Brief Title: A Study to Investigate the Treatment Effect of Subcutaneous Injections of Pentosan Polysulfate Sodium Compared With Placebo in Adult Participants With Knee Osteoarthritis Pain.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Paradigm Biopharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PARA_OA_012
Record Dates: First submitted 2025-03-11; First posted 2025-04-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PPS (Active Comparator): Pentosan polysulfate sodium 2mg/kg twice weekly for 6 weeks
  Interventions: Drug: Pentosan Polysulfate Sodium twice weekly
- Placebo (Placebo Comparator): Placebo (Sodium Chloride Injection, 0.9%) twice weekly for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentosan Polysulfate Sodium twice weekly — Subcutaneous injection, 2 mg/kg twice weekly for 6 weeks
  Arms: PPS
Drug: Placebo — Placebo, subcutaneous injection, twice weekly for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the change in pain and function with subcutaneous injections of pentosan polysulfate sodium (PPS) compared with subcutaneous injections of placebo in participants with knee OA pain.

Study details include:

* The study duration will be up to 64 weeks.
* The treatment duration will be 6 weeks.
* The visit frequency will be twice weekly during treatment.
* The visit/contact frequency will be every 4-6 weeks during the 52-week Follow-up period.
* Approximately 466 participants will be enrolled into this study.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, multicenter study that will evaluate the dose and treatment effect of PPS in participants with knee OA pain.

Participants will be randomised 1:1 to receive twice-weekly subcutaneous (SC) injections of 2 mg/kg PPS or placebo for 6 weeks.

An interim analysis for a potential early conclusion is planned after approximately 50% of participants complete Day 112.

The primary analysis will be conducted when all participants complete Day 112. A final analysis will be conducted when the last participant reaches Day 404.

The maximum duration for each participant is up to 64 weeks, which includes

* 7-week Screening Period from Day -45 to Day -1
* 6-week Treatment Period from Day 1 to Day 39
* 52-week Follow-up Period from Day 40 to Day 404

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 years of age inclusive, at the time of signing the informed consent.
2. Clinical diagnosis of OA in the index knee by American College of Rheumatology 1986 criteria.
3. Radiographic diagnosis (confirmed by radiologist) of knee OA classified K-L grade 2, 3, or 4 on standing anterior-posterior X-ray of the index knee.
4. Participant is unresponsive for at least 6 months preceding Screening to any two combinations of OA therapies (one from each A and B) within the last 12 months that include: A.) conservative non-pharmacologic therapy (exercise, weight loss, physical therapy) or simple analgesics (e.g., acetaminophen) and B.) pharmacological treatment (topical or oral NSAIDs [or cyclooxygenase (COX) inhibitor], or intra-articular [IA] injections), or participant is unable to take NSAIDs because of contraindication or inability to tolerate.
5. Average daily pain (ADP) numerical rating scale (NRS) score of 4-9 in the index knee at Screening.
6. Baseline average weekly ADP NRS score of 4-9 in the index knee in the 7 days prior to randomization.
7. No more than one 24-hr average pain score (0-10 NRS) reported as "10" during the 7 days prior to Day 1.
8. Body mass index of ≥18.0 to ≤39.0 kg/m2.
9. Female subjects of childbearing potential and Male subjects must agree to comply with protocol specified contraceptive requirements
10. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
11. Completion of at least 11 out of 14 ADP NRS scores for at least 14 days prior to randomisation.
12. Current non-pharmacologic treatment regimen for knee OA (excluding knee brace) must be stable for at least 2 weeks before Day 1 and remain stable throughout the study. Participant must be willing to abstain from starting a new or changing their non-pharmacologic treatment regimen for the duration of the study.
13. Willing to stop treatment with oral and topical NSAIDs, and all other systemic pain medications (except allowed rescue medication) from 2 weeks before Day 1 to end of study.
14. Agrees to use acetaminophen/paracetamol or topical analgesics (topical NSAIDs are prohibited) as rescue therapy if required.

Exclusion Criteria:

1. History of idiopathic or immune-mediated thrombocytopenia including history of HIT with or without thrombosis.
2. History of major bleeding disorders including haemophilia.
3. Currently active or recent history (within preceding 12 months) of a gastric or duodenal ulcer, or suspicion of gastrointestinal tract bleeding.
4. Recent cerebral bleeding or operation on brain, spine, or eyes within 12 months of Day 1.
5. Spinal anaesthesia within 14 days of Day 1.
6. Fibromyalgia, regional pain caused by lumbar or cervical compression with radiculopathy, or other moderate to severe pain disorder that may confound assessments or self-evaluation of the pain associated with osteoarthritis. Participants with a present (current) history of sciatica are not eligible for participation. Participants with a history of sciatica who have been asymptomatic for ≥3 months and who have no evidence of radiculopathy or sciatic neuropathy on thorough neurologic examination are eligible for participation.
7. History of other disease that may involve the index knee, including inflammatory joint disease such as rheumatoid arthritis (RA), seronegative spondyloarthropathy (e.g., ankylosing spondylitis, psoriatic arthritis, inflammatory bowel disease-related arthropathy), crystalline disease (e.g., gout), endocrinopathies, metabolic joint diseases, lupus erythematosus, joint infections, Paget's disease, or tumours.
8. History of hypersensitivity to PPS, heparin or heparin-like drugs, or drugs of a similar chemical or pharmacological class.
9. Predisposition to hypersensitivity due to multiple (2 or more) atopic diseases (such as atopic eczema, asthma, and chronic allergic rhinitis and/or rhinoconjunctivitis) or multiple (2 or more) severe allergies.
10. Allergy or contraindication to tetracosactide (Synacthen®), cosyntropin (Cortrosyn®).
11. Allergy or contraindication to gadolinium.
12. Chronic medical conditions including but not limited to those stated below requiring medical regime changes within 60 days before Day 1.

    Concurrent unstable peripheral, cardiac, and cerebral vascular disease, poorly controlled chronic obstructive pulmonary disease and asthma, coagulopathies, uncontrolled neurological conditions, active tuberculosis, active infections, symptomatic cardiac arrhythmias, adrenal insufficiency (primary or central), nephrotic syndrome, cirrhosis (Child-Pugh stage B or C), Gilbert syndrome, uncontrolled diabetes, and uncontrolled hypothyroidism or hyperthyroidism, or mental or emotional disorders that preclude reliable study participation.
13. History of pituitary irradiation or recent (within 1 year) history of transsphenoidal surgery.
14. Any cancer within the previous 5 years, except for basal cell carcinomas.
15. History or current autoimmune polyglandular syndromes.
16. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per the protocol.
17. Current treatment with anticoagulants or antiplatelet drugs within 2 weeks before Day 1, excluding aspirin ≤150 mg/day.
18. Previous treatment with PPS in any form.
19. Current or recent (within 90 days before Day 1) immunosuppressive or immunomodulatory (with immunosuppressive effects) systemic therapy including but not limited to oral, inhaled, intranasal, intra-articular (IA) and topical corticosteroids (occasional use of topical, inhaled or intranasal corticosteroids is acceptable).
20. Use of NSAIDs with 2 weeks before Day 1.
21. Use of opioids within 6 weeks before Day 1.
22. Use of glucosamine or chondroitin within 6 weeks before Day 1.
23. Use of bisphosphonates and denosumab within 12 weeks before Day 1.
24. Use of iloprost within 12 weeks before Day 1.
25. Use of a knee brace on the index knee within 2 weeks before Day 1.
26. Systemic steroids administered intravenously, intramuscularly, or orally for OA or other indications within 8 weeks before Day 1.
27. Intra-articular (IA) injections to the index knee: steroids within 12 weeks before Day 1; hyaluronic acid (HA) or any other IA injections within 24 weeks before Day 1.
28. Stem cells or platelet-rich plasma within 12 months of Day 1.
29. Cannabinoids within 30 days before Day 1.
30. Use of individual vitamins and dietary supplements known to alter haemostasis within 2 weeks before Day 1, including ajoene, birch bark, cayenne, Chinese black tree fungus, cumin, evening primrose oil, feverfew, garlic, ginger, ginkgo biloba, ginseng, grapeseed extract, milk thistle, omega 3 fatty acids, onion extract, St. John's wort, turmeric, vitamins C and E, vitamin K, (multivitamins allowed).
31. Known exposure to heparin within the last 100 days as determined by history of drug use or history of the following medical conditions or interventions: cardiac bypass surgery or thromboembolic disease.
32. Treatment with dehydroepiandrosterone sulfates (DHEA-S) within 6 weeks before Day 1.
33. Chronic use of oral glucocorticoid receptor antagonists or cortisol synthesis inhibitors within 12 weeks before Day 1.
34. Biotin within 72 hours before Screening.
35. Megestrol acetate within 6 weeks before Day 1.
36. Participation in another clinical trial or administration of any IP or experimental product within 24 weeks or 5 half-lives (whichever is longer) before Day 1.
37. Activated partial thromboplastin time [aPTT]) > 36 seconds, platelets <150,000/μL, or liver enzyme tests (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) ≥ 2 × ULN at Screening.
38. Total bilirubin ≥1.5 ULN.
39. Active or chronic hepatitis B virus, hepatitis C virus, or uncontrolled HIV infection (detectable virus or diagnosis of AIDS); participants with HIV infection must be on chronic suppressive antiviral medication.
40. Evidence of any of the following conditions in any screening imaging: excessive malalignment (≥10 degrees varus or valgus) of the knee, subchondral insufficiency fracture (SIF), osteonecrosis/bone infarct, osteochondritis dissecans, stress or acute fracture, atrophic OA, pathologic fracture, primary or metastatic tumour, infectious arthritis or osteomyelitis, chronic or acute, Charcot's knee joint, synovial chondromatosis, certain posterior root tears of the meniscus, bone contusion, bone marrow oedema syndrome, bone marrow infiltration, gout, severe chondrocalcinosis, other arthropathies (e.g., RA, psoriatic arthritis), systemic metabolic bone disease (e.g., Paget's disease, metastatic calcifications) or other conditions identified by a radiologist or Medical Monitor which may interfere with a participant's assessment of pain.
41. Any clinically significant abnormalities on clinical chemistry, haematology, urinalysis, physical examination, medical history, or vital signs as judged by the Investigator (at Screening).
42. Resting, supine blood pressure (BP) ≥160 mmHg in systolic pressure or ≥100 mmHg in diastolic pressure at Screening. If a participant is found to have uncontrolled and/or untreated significant hypertension at Screening and antihypertensive treatment is initiated, assessment for study eligibility should be deferred until BP and antihypertensive medication have been stable for at least 1 month. For participants with previously diagnosed hypertension, antihypertensive medications must be stable for at least 1 month before Screening.
43. Any macular findings on clinical examination or imaging suggestive of: moderate or advanced dry macular degeneration, geographic atrophy, moderate or advanced myopic degeneration, wet macular degeneration, pattern dystrophy or other pigmentary maculopathy, moderate or severe diabetic or hypertensive retinopathy, recent retinal vascular occlusion, macular hole or advanced epiretinal membrane with associated macular oedema, retinal dystrophy, toxic retinal maculopathy, chronic central serous retinopathy, presence of significant subretinal or intraretinal fluid (OCT finding), presence of vitelliform or vitelliform-like macular changes (OCT and clinical finding), severe maculopathy not otherwise specified.
44. Morning cortisol <3 μg/dL.
45. Adrenocorticotropic hormone (ACTH) <10 pg/mL.
46. US/Canada only: Morning cortisol ≥3 μg/dL and <10 μg/dL and peak cortisol (by ACTH stimulation [250 μg, IM] test) <18 μg/dL at both 30 min and 60 min post stimulation.
47. Current hyperkalaemia and/or hyponatremia.
48. Contraindication to MRI.
49. Largely or wholly incapacitated (e.g., bedridden or confined to a wheelchair, permitting little or no self-care).
50. Major surgery or anticipated surgery during the study.
51. Currently hospitalised or any planned hospitalizations during the study.
52. Plan for total knee reconstruction in affected knee(s) during the study.
53. Knee surgery or trauma to the index knee within 1 year before Day 1.
54. A history of drug or alcohol abuse and/or dependence within the 12 months before Screening that, in the opinion of the Investigator, may affect participant ability to comply with study requirements.
55. An employee of the Sponsor, clinical research organisation(s), or research site personnel directly affiliated with this study or their immediate family members defined as a spouse, parent, sibling, or child, whether biological or legally adopted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at Day 112 in knee pain as assessed by the weekly average of daily pain (ADP) score on the numerical rating scale (NRS) 11-point (0-10) scale. | Baseline, Daily to Day 112
  The NRS is an 11-point unidimensional scale for self-report of pain. The participant selects a whole number (0-10) that best reflects the intensity of their pain. The anchors are 0=no pain and 10=extreme pain/worst possible pain. It is often categorised into no pain=0, mild pain=1-3, moderate pain=4-6, severe pain=7-10.
  Participants will be asked to consider their average pain over the last 24 hours.

SECONDARY OUTCOMES:
Change from baseline in function as assessed by the average functional subscale score of the WOMAC NRS 3.1 Index | Measured at 20 timepoints from Day 1 to 404.
  The WOMAC NRS 3.1 Index is a validated, self-administered, health status questionnaire that assesses pain, stiffness, and function in patients with hip or knee OA (Bellamy et al., 1988).
  The WOMAC NRS 3.1 Index consists of 24 questions and produces 3 subscale scores for pain (5 questions), stiffness (2 questions), and function (17 questions) and a total score that summarises overall disability. Each question is scored from 0 to 10 using a standardised 11-point NRS.
  Each subscale score and the total score will be averaged to provide subscale and total scores between 0 and 10.
  Participants are to consider their last 4 hours when answering the questions.
Change from baseline in knee pain as assessed by the average pain subscale score of the WOMAC NRS 3.1 Index | Measured at 20 timepoints from Day 1 to 404.
  The WOMAC NRS 3.1 Index is a validated, self-administered, health status questionnaire that assesses pain, stiffness, and function in patients with hip or knee OA (Bellamy et al., 1988).
  The WOMAC NRS 3.1 Index consists of 24 questions and produces 3 subscale scores for pain (5 questions), stiffness (2 questions), and function (17 questions) and a total score that summarises overall disability. Each question is scored from 0 to 10 using a standardised 11-point NRS.
  Each subscale score and the total score will be averaged to provide subscale and total scores between 0 and 10.
  Participants are to consider their last 4 hours when answering the questions.
Change from baseline in knee pain as assessed by the weekly average of daily pain (ADP) score on the numerical rating scale (NRS) 11-point (0-10) scale. | Measured at 21 timepoints from Screening to Day 404.
  The NRS is an 11-point unidimensional scale for self-report of pain. The participant selects a whole number (0-10) that best reflects the intensity of their pain. The anchors are 0=no pain and 10=extreme pain/worst possible pain. It is often categorised into no pain=0, mild pain=1-3, moderate pain=4-6, severe pain=7-10.
  Participants will be asked to consider their average pain over the last 24 hours.
Change from baseline in Patient Global Impression of Change (PGIC) | Measured at 10 timepoints from Days 39 to 404.
  The PGIC is a self-administered question that rates participants' overall improvement in chronic pain since beginning treatment from 1 "no change (or condition has worsened)" to 7 "a great deal better" in response to the question "Since beginning treatment, how would you describe the change (if any) in activity, limitation, symptoms, emotions, and overall QoL related to your arthritis".
Change from baseline in knee stiffness as assessed by the average stiffness subscale score of the WOMAC NRS 3.1 Index | Measured at 20 timepoints from Day 1 to 404.
  The WOMAC NRS 3.1 Index is a validated, self-administered, health status questionnaire that assesses pain, stiffness, and function in patients with hip or knee OA (Bellamy et al., 1988).
  The WOMAC NRS 3.1 Index consists of 24 questions and produces 3 subscale scores for pain (5 questions), stiffness (2 questions), and function (17 questions) and a total score that summarises overall disability. Each question is scored from 0 to 10 using a standardised 11-point NRS.
  Each subscale score and the total score will be averaged to provide subscale and total scores between 0 and 10.
  Participants are to consider their last 4 hours when answering the questions.
Change from baseline overall as assessed by the overall score of the WOMAC NRS 3.1 Index | Measured at 20 timepoints from Day 1 to 404.
  The WOMAC NRS 3.1 Index is a validated, self-administered, health status questionnaire that assesses pain, stiffness, and function in patients with hip or knee OA (Bellamy et al., 1988).
  The WOMAC NRS 3.1 Index consists of 24 questions and produces 3 subscale scores for pain (5 questions), stiffness (2 questions), and function (17 questions) and a total score that summarises overall disability. Each question is scored from 0 to 10 using a standardised 11-point NRS.
  Each subscale score and the total score will be averaged to provide subscale and total scores between 0 and 10.
  Participants are to consider their last 4 hours when answering the questions.
Proportion of participants with ≥30% and ≥50% pain reduction from baseline as assessed by the average pain subscale score of the WOMAC NRS 3.1 Index. | Measured at 20 timepoints from Day 1 to 404.
  The WOMAC NRS 3.1 Index is a validated, self-administered, health status questionnaire that assesses pain, stiffness, and function in patients with hip or knee OA (Bellamy et al., 1988).
  The WOMAC NRS 3.1 Index consists of 24 questions and produces 3 subscale scores for pain (5 questions), stiffness (2 questions), and function (17 questions) and a total score that summarises overall disability. Each question is scored from 0 to 10 using a standardised 11-point NRS.
  Each subscale score and the total score will be averaged to provide subscale and total scores between 0 and 10.
  Participants are to consider their last 4 hours when answering the questions.
Proportion of participants with ≥30% and ≥50% improvement in function from baseline as assessed by the average pain subscale score of the WOMAC NRS 3.1 Index. | Measured at 20 timepoints from Day 1 to 404.
  The WOMAC NRS 3.1 Index is a validated, self-administered, health status questionnaire that assesses pain, stiffness, and function in patients with hip or knee OA (Bellamy et al., 1988).
  The WOMAC NRS 3.1 Index consists of 24 questions and produces 3 subscale scores for pain (5 questions), stiffness (2 questions), and function (17 questions) and a total score that summarises overall disability. Each question is scored from 0 to 10 using a standardised 11-point NRS.
  Each subscale score and the total score will be averaged to provide subscale and total scores between 0 and 10.
  Participants are to consider their last 4 hours when answering the questions.
Number of days of rescue medication used | Recorded from Day 1 to 404
  In case of inadequate pain relief, either acetaminophen/paracetamol up to 3000 mg per day or topical analgesics, up to 4 days in a week may be taken as rescue medication between day 1 and Day 404. Participants will record all use of rescue and other pain medications/therapies in their electronic diary.
Change from baseline in QoL as assessed by EQ-5D-5L. | Measured at 13 timepoints from Days 1 to 404
  The EQ-5D-5L questionnaire is a self-assessed, health related, QoL questionnaire consisting of the EQ-5D descriptive system and the EQ VAS. The descriptive system comprises of five dimensions, where each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions.
Change from baseline in cartilage volume and thickness on Magnetic Resonance Imaging (MRI). | Measured at Days 1, 168 and 404.
  Gadolinium MRI images will be taken to measure changes in cartilage volume and thickness.
Change from baseline in joint synovitis/effusion volume on Magnetic Resonance Imaging (MRI). | Measured at Days 1, 168 and 404.
  Gadolinium MRI images will be taken to measure changes in joint synovitis/effusion volume,.
Change from baseline in subchondral BML area and volume on Magnetic Resonance Imaging (MRI). | Measured at Days 1, 168 and 404.
  Gadolinium MRI images will be taken to measure changes in subchondral BML area and volume,.
Change from baseline in bone shape/osteophytes on Magnetic Resonance Imaging (MRI). | Measured at Days 1, 168 and 404.
  Gadolinium MRI images will be taken to measure changes in bone shape/osteophytes.
Change from baseline in joint space width on X-ray. | Measured at Days 1 and 404.
  X-ray for comparison of joint space width
OMERACT-OARSI Responder Index response rate | Measured at 10 timepoints from Days 39 to 404.
  OMERACT-OARSI-Outcome Measures in Rheumatology-Osteoarthritis Research Society International.
  Participants are considered as an OMERACT-OARSI responder: if the change (improvement) from baseline to day of interest was greater than or equal to >= 50 percent and >= 2 units in either WOMAC pain sub-scale or physical function sub-scale score; if change (improvement) from baseline to week of interest was >=20 percent and >=1 unit in at least 2 of the following: 1) WOMAC pain sub-scale score, 2) WOMAC physical function sub-scale score, 3) Patient Global Impression of Change (PGIC).
Change from baseline in Work Productivity and Activity Impairment (WPAI) questionnaire score | Measured at 10 timepoints from Day 39 to 404.
  The WPAI questionnaire (WPAI:OA-knee) is a validated self-administered questionnaire that assesses work impairment due to OA . The questionnaire gathers information on employment status, hours worked, hours missed due to OA, and hours missed for any other reasons.
Incidence of treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs) | From enrollment to Day 404
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
  An SAE is any untoward medical occurrence that at any dose results in one or more of the following outcomes: death; life-threatening; requires in-patient hospitalization or prolongation of an existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; is an important medical event.
  Treatment-emergent means events occurring between the first dose of study drug and up to Day 404 that were absent before treatment or that worsened relative to pre-treatment state.
Incidence of treatment-emergent clinical abnormalities | From enrollment to Day 404
  Treatment-emergent clinical laboratory abnormalities are abnormalities in laboratory results between the first dose of study drug and up to Day 404 that were absent before treatment or that worsened relative to pre-treatment state

OTHER OUTCOMES:
Exploratory: Characterize the AUC profile of single and multiple doses based on sparse blood sampling. (pharmacokinetic subset only) | Days 1, 15 and 39 - pre-dose and 2, 4, and 6 hours. Pre-dose on day 4, 8, 11, 18, 22, 25, 29, 32, 36 and 39
  Blood samples for assay of plasma PPS concentration will be obtained from a subset of patients before dosing and 2, 4, and 6 hours after dosing on study Days 1, 15 and 39. On other days, a pre-dose sample will be collected. Samples will be assayed using a sensitive, validated bioanalytical method.
  Plasma concentrations of PPS will be tabulated by time and participant and inspected for relationship to dose during titration and stable treatment phases.
Exporatory: Number of participants with an Anti-Drug-Antibody (ADA) response after treatment and correlation with clinical events. | Baseline, Days 11, 25, 39, 56 and 84.
  Human serum ADA samples will be analyzed for the presence or absence of anti-drug-antibodies by using a semi-quantitative enzyme linked immunosorbent assay (ELISA).
Exploratory: Change from baseline in serum biomarkers, including but not limited to, COMP, aggrecan ARGS, CRTAC-1, PRO-C2 PIIBNP, NTx-Ⅰ, and HA. | Measured at 11 timepoints from Day 4 to 168.
  ARGS-(aggrecan) alanine-arginine-glycine-serine; COMP-cartilage oligomeric matrix protein; CRTAC-1-cartilage acidic protein-1; HA-hyaluronic acid; NTx-1-N-terminal telopeptide of type I collagen; PIIBNP-N-terminal propeptide of type II collagen; PRO-C2-type II collagen C-terminal propeptide.
Exploratory: Change from baseline of cartilage volume and thickness and whether these correlate with clinical pain outcomes. | Screening, Day 168 and 404
  The correlation co-efficient of changes in cartilage volume and thickness as measured on MRI and pain clinical outcomes.
Exploratory: Change from baseline of subchondral BMLs, and whether these correlate with clinical pain outcomes. | Screening , Day 168 and 404
  The correlation co-efficient of changes in subchondral BMLs as measured on MRI and pain clinical outcomes.
Exploratory: Change from baseline of bone shape and whether these correlate with clinical pain outcomes. | Screening , Day 168 and 404
  • The correlation co-efficient of changes in bone shape changes as measured on MRI and pain clinical outcomes
Exploratory: Change from baseline of joint space width and whether these correlate with clinical pain outcomes. | Screening and 404
  The correlation co-efficient between changes in joint space width as measured on X-Ray and clinical pain outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Medical, Study Director — Paradigm Biopharmaceuticals
Locations (34):
- United States (27):
  - Onyx Clinical Research-Peoria, Peoria, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Orange County Research Institute, Anaheim, California
  - Core Healthcare Group, Cerritos, California
  - Arrow Clinical Trials, Daytona Beach, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Well Pharma Medical Research, Miami, Florida
  - K2 Medical Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Phoenix Clinical Research, Tamarac, Florida
  - Conquest Research, Winter Park, Florida
  - Chicago Clinical Research, Inc, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Profound Research, Farmington Hills, Michigan
  - Insight Research Institute, Flint, Michigan
  - Rochester Medical Group, Rochester Hills, Michigan
  - Onyx Clinical Research - Rochester Hills, Troy, Michigan
  - Physician Research Collaboration, Lincoln, Nebraska
  - Drug Trials America, Hartsdale, New York
  - IMC Clinical Research Manhattan, New York, New York
  - FutureSearch Trials of Neurology, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Vilo Research Group, Houston, Texas
  - DM Clinical Research, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Quality Research Inc., San Antonio, Texas
- Australia (7):
  - Canopy Clinical Research-Northern Beaches, Brookvale, New South Wales
  - Novatrials, Charlestown, New South Wales
  - Canopy Clinical Research-Wollongong, Wollongong, New South Wales
  - Mater Health Brisbane, South Brisbane, Queensland
  - Griffith University, Southport, Queensland
  - Sportsmed, Stepney, South Australia
  - Sportsmed Biologic LTD, Box Hill, Victoria

IPD SHARING:
Plan to Share IPD: No